CLINICAL TRIAL: NCT03204266
Title: Oral Supplementation to Enhance Recovery Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0117; NCI-2018-01132 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Malignant Neoplasms of Urinary Tract
Keywords: urinary tract; Bladder cancer; Radical cystectomy; Omega-3 Fatty Acids
MeSH Terms: conditions — Urologic Neoplasms; Urinary Bladder Neoplasms | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immunonutrition: ARS + Omega-3 Fatty Acids (Experimental): Participants take 1 ounce (30mls) of Arginine recovery supplement (ARS) four times daily 5 days preoperatively and 14 days postoperatively.
  Participants also given omega-3 fatty acids, 1 gram four times a day, 4 grams total per day. This will be started 7 days preoperatively and continued 14 days postoperatively.
  Interventions: Drug: Arginine recovery supplement; Dietary Supplement: Omega-3 Fatty Acids
- No Immunonutrition (No Intervention): Participants receive regular enhanced recovery after surgery (ERAS)/Optimized Surgical Journey (OSJ) education and follow up.

INTERVENTIONS:
Drug: Arginine recovery supplement — Participants take 1 ounce (30mls) of Arginine recovery supplement four times daily 5 days preoperatively and 14 days postoperatively.
  Other Names: ARS
  Arms: Immunonutrition: ARS + Omega-3 Fatty Acids
Dietary Supplement: Omega-3 Fatty Acids — Participants given omega-3 fatty acids, 1 gram four times a day, 4 grams total per day. This will be started 7 days preoperatively and continued 14 days postoperatively.
  Arms: Immunonutrition: ARS + Omega-3 Fatty Acids

SUMMARY:
The goal of this clinical research study is to learn the supplements Pro-Stat (which has l-arginine and also contains protein) and omega-3 fatty acids will be well tolerated in patients who have radical cystectomy for bladder cancer. Researchers also want to learn how these medications affect inflammation and recovery for these surgical patients.

This is an investigational study. Pro-Stat is not FDA-approved to treat any specific condition or disease. Omega-3 fatty acids are FDA-approved to treat high triglyceride levels. Their use to treat inflammation and help improve recovery after bladder cancer surgery is investigational.

The study doctor can explain how the supplements are designed to work.

Up to 46 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to perform a few tasks to learn about your strength, memory, and nutrition. These should take about 20 minutes to complete.

Study Groups:

You will be randomly assigned (as in the flip of a coin) into 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If you are in Group 1, you will receive the Pro-Stat and omega-3 fatty acid supplements.
* If you are in Group 2, you will not receive the Pro-Stat and omega-3 fatty acid supplements.

You will be asked to write down any supplements you take in a diary that will be provided to you. You should write down any supplements you take for the week before and 2 weeks after surgery. Please bring this diary to your follow up appointment after surgery.

Supplement Administration:

If you are in Group 1, you will receive the omega-3 fatty acids in a pill bottle and the Pro-Stat in foil packets. You should take each supplement 4 times daily. Omega-3 fatty acid capsules should be swallowed whole and should not be opened, chewed, or crushed.

Packets of Pro-Stat may be mixed with other liquids or food. If vomiting occurs, do not replace the vomited dose. If you miss a dose, you may take an extra dose that same day.

You should bring all supplements you haven't taken with you to your 14 day visit after surgery.

Length of Study Participation:

Your doctor may lower the dose of the supplements if you experience any serious side effects that may be related to the supplements. If these side effects continue after the dose has been lowered, you will no longer be able to take the supplements. You may also be taken off study if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Surgery:

You will have your standard-of-care surgery. You will receive a separate consent for the surgery that explains the procedure and the risks.

Study/Follow-Up Visits:

Before Surgery:

* Blood (about 8 teaspoons) will be drawn for routine tests, protein testing, biomarker testing, to check your cholesterol, liver function, your amino acid levels, and to test for inflammatory markers. Biomarkers are found in the blood and may be related to your reaction to the supplements.
* Urine will be collected for routine tests.
* Blood (about 4 teaspoons) will also be drawn and stored at MD Anderson for future testing as a part of this study.

Day 1 After Surgery:

* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 4 teaspoons) will also be drawn and stored at MD Anderson for future testing as a part of this study.

Day 2 After Surgery, blood (about 2 teaspoons) will be drawn for routine tests.

Day 3 After Surgery:

* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 4 teaspoons) will also be drawn and stored at MD Anderson for future testing as a part of this study.

On your Day of Discharge from the hospital:

* Blood (about 2 teaspoons) will be drawn for routine tests.
* Urine will be collected for routine tests.

Day 14 After Surgery:

* Blood (about 2 teaspoons) will be drawn for routine tests, to check your cholesterol, your liver function, and your amino acid levels.
* Urine will be collected for routine tests.
* Blood (about 4 teaspoons) will also be drawn and stored at MD Anderson for future testing as a part of this study.

You weight will be measured at all of the above visits and information will be collected from your medical record.

Day 90 After Surgery, you will have a physical exam and your weight will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing RC for bladder cancer with urinary diversion at MD Anderson Cancer Center (MDACC). All races and ethnicities will be included
2. Patients must be willing to spend time for the study
3. Patient must provide signed informed consent.
4. Male or female, age >/= 18 years.
5. Adequate hepatic function: alkaline phosphatase </= 1.5 x Upper Limit of Normal (ULN); total bilirubin, aspartate aminotransferase (AST), and Alanine aminotransferase (ALT) </= 1.5 x ULN; international normalized ratio (INR) <1.3 (or <3 if on anticoagulant therapy).

Exclusion Criteria:

1. Subjects will be excluded if they do not attend pre-operative clinic dedicated to RC subjects.
2. Subjects with allergies to any supplements.
3. Subjects with galactosemia will be excluded.
4. Subjects may be excluded if they have known autoimmune inflammatory disease. (e.g. rheumatoid arthritis, ulcerative colitis, gout, chronic steroids).
5. Hepatic impairment: alkaline phosphate > 1.5 x ULN; total bilirubin, AST, and ALT > 1.5 x ULN; INR >1.3 (or >3 if on anticoagulant therapy).
6. Previously unable to tolerate either supplement due to taste or gastrointestinal (GI) side effects.
7. Any active malignancies being treated other than bladder cancer (incidentally found prostate cancer at RC is acceptable).
8. Unwillingness or inability to comply with mandated blood draws.
9. Any previous immunotherapy with immune checkpoint inhibitors such was Nivolumab, Atezolizumab and others in the class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Determination if novel immunonutrition regimen is able to be implemented with adequate compliance in Radical Cystectomy (RC) patients: Participant Compliance | 21 days after starting immunonutrition regimen
  Participant compliance defined as "Yes" if a participant completes at least 16 out of the total 21 days' treatment.

SECONDARY OUTCOMES:
Determination if Poor Recovery is Associated With the Use Immunonutrition Before and After Radical Cystectomy (RC): Length of Hospital Stay>7 Days | 90 days after surgery
  Poor recovery determined by length of stay greater than 7 days.
Determination if Poor Recovery is Associated With the Use Immunonutrition Before and After Radical Cystectomy (RC): Postoperative Infections | 90 days after surgery
  Poor recovery determined by any postoperative infection.
Determination if Poor Recovery is Associated With the Use Immunonutrition Before and After Radical Cystectomy (RC): Hospital Readmissions | 90 days after surgery
  Poor recovery determined by hospital readmission within 90 days after radical cystectomy.
Determination if Poor Recovery is Associated With the Use Immunonutrition Before and After Radical Cystectomy (RC): Deaths within 90 days of Cystectomy | 90 days after surgery
  Poor recovery determined by death within 90 days of cystectomy.
Decrease in Inflammatory Response of Serum Interleukin-6 Levels After Radical Cystectomy (RC) postoperative day 1 | 1 day after surgery
  IL-6 levels drawn postoperative day 1 within 24 hours of anesthesia induction. This used to create a response curve based on the administration of immunonutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Neema Navai, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org